CLINICAL TRIAL: NCT04486287
Title: Phase II Study of PD-1 Inhibitor With Sintilimab After Stereotactic Ablation Brachytherapy for Refractory Oligometastatic Non-Small Cell Lung Cancer
Brief Title: Sintilimab After Stereotactic Ablation Brachytherapy for Refractory Oligometastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA-SABT
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Oligometastasis; Lung Neoplasms
Keywords: PD-1 inhibitor,Brachytherapy,SABT,Oligometastatic,NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab Arm (Experimental): Sintilimab after Stereotactic Ablation Brachytherapy.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg IV, every 3 weeks, until progressive disease (PD), intolerable toxicity, or at a maximum of 12 months.
  Before enrollment, patient should undergo Stereotactic Ablation Brachytherapy. Sintilimab shall be started no later than 4 weeks after Stereotactic Ablation Brachytherapy.
  Other Names: Tyvyt; IBI 308

SUMMARY:
The study aim to investigator the efficacy and safety of sintilimab after Stereotactic Ablation Brachytherapy(SABT) for refractory oligometastatic non-small cell lung cancer(NSCLC), who had failed second-line systemic therapy.

DETAILED DESCRIPTION:
This study is a single-arm phase II study of sintilimab after SABT for refractory oligometastatic NSCLC, who had failed second-line systemic therapy.In this study, 44 patients with oligometastatic NSCLC were treated with sintilimab after SABT every 3 weeks until disease progression and intolerance. Toxicity, withdrawal of informed consent, death or other cessation of treatment as prescribed by the program, whichever occurs first. The primary end point was the ORR based on RECIS 1.1, which was evaluated by the Independent Imaging Review Board (IRRC). An interim analysis will be conducted during the course of the study. The results and reports will be provided to the Independent Data Audit Committee (IDMC), which determines whether the trial is valid based on the valid cut-off value of the trial and whether the study data can be submitted in advance. Make recommendations to the sponsor. Prior to the interim analysis, the IDMC charter will be finalized and approved by IDMC and the sponsor. The responsibilities and related procedures of IDMC members will be defined in the IDMC charter.

ELIGIBILITY:
Inclusion Criteria:

1.Provide written informed consent for the trial.

2.18 years of age on day of signing informed consent.

3.Completion of definitive therapy 4-12 weeks prior to enrollment. There are no specific limitations on which treatment modalities can be used in the definitive setting (e.g. the use of adjuvant chemotherapy is acceptable), but all other treatments must be complete at least 4 weeks prior to enrollment.

4.Patients confirmed by histological specimens who are not eligible for EGFR, ALK or ROS1 targeted therapy (with no tumor) EGFR-sensitive mutations and no evidence of ALK, ROS1 gene rearrangement.

5.Patients must have disease progression or recurrence after receiving first line systemic therapy for advanced or metastasis disease: 1) Maintenance therapy after platinum based chemo-doublet shall not be considered as a separated treatment regimen, 2)Patients who had received neo-adjuvant/adjuvant therapy or radical chemo- radiotherapy for local advanced disease and relapsed after 6 month or later, must have failed second-line treatment for recurrent disease before enrollment.

6.ECOG PS 0-2, with expected survival over 3 months.

7.Adequate hematopoietic function, defined as: absolute neutrophil count (ANC) ≥ 1.5 x 10*9/L; platelet count ≥100 x 10*9/L; hemoglobin ≥90 g/L [no blood transfusion within 7 days or not erythropoietin (EPO) dependent].

8.Adequate liver function, defined as: total serum bilirubin ≤ 1.5 x upper limit of normal (ULN); serum alanine transaminase (ALT) and aspartic transaminase (AST) ≤ 2.5 x ULN, with no liver transplantation.

9.Adequate renal function, defined as: serum creatinine ≤ 1.5 x ULN or calculated creatinine-clearance ≥ 60 ml/min (Cockcroft-Gault). Urine protein less than 2+ by urinalysis or 24-hour urinary protein quantity < 1g.

10.Adequate coagulation function, defined as: international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN. For patients receiving anticoagulant therapy can be enrolled if PT is within the range defined by anticoagulant therapy.

11.Myocardial enzymes are within normal range.

12.For all female patients of childbearing potential, a negative pregnancy test (either urine or serum) must be obtained within 3 days before the first dose (Cycle 1, Day 1) of study treatment. If a urine pregnancy test shows an unconfirmed result, a serum pregnancy test must be performed.

13.All subjects of childbearing potential must agree to use efficient contraceptive methods that result in a failure rate of < 1% per year during the study treatment period and for at least 180 days after discontinuation from study treatment.

Exclusion Criteria:

1. Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Diagnosis of immunodeficiency or exposure to systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (Nasal or oral inhalers are permissible).
3. Prior monoclonal antibody within 4 weeks prior to study Day 1 or individuals who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Day 1 drug administration on study or inability to recover (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
5. Note: Subjects with ≤ Grade 2 neuropathy or alopecia are exceptions to this criterion and may qualify for the study.
6. Note: If subject had major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Known additional malignancy that is progressing or requires active treatment.
8. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, non-invasive bladder tumors, or in situ cervical cancer
9. Known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis.
10. Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule.Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome are not excluded from the study.
11. Evidence of pre-existing interstitial lung disease or active, non-infectious pneumonitis.
12. Active infection requiring systemic therapy with IV antibiotics
13. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
17. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Known active Hepatitis B (e.g., HBsAg positive or HBV DNA detectable) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Receipt of live vaccine within 30 days prior to the first dose of trial treatment.
20. Progressive disease or sites of new metastasis after definitive therapy for oligometastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months after enrollment or study close.
  ORR(RECIST 1.1 as assessed by the investigator )is defined as the proportion of patients with a complete response (CR) or partial response (PR) as their best response.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months after enrollment or study close.
  Time to progression or death from initiation of Stereotactic Ablation Brachytherapy.
Overall Survival(OS) | up to 24 months after enrollment or study close.
  Defined as the time until death due to any cause.
Disease Control Rate (DCR) | up to 24 months after enrollment or study close .
  RECIST 1.1 as assessed by the investigator) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD).
Treatment-related Adverse Events (AEs) | From the date of randomization to 90 days after last dose of study treatment .
  Evaluation of adverse event rate according to CTCAE(Common terminology criteria for adverse events) v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: BIN HUO, Principal Investigator — Tianjin Medical Unversity Second Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergsma DP, Salama JK, Singh DP, Chmura SJ, Milano MT. Radiotherapy for Oligometastatic Lung Cancer. Front Oncol. 2017 Sep 19;7:210. doi: 10.3389/fonc.2017.00210. eCollection 2017. PMID 28975081
- [Background] Gong HY, Wang Y, Han G, Song QB. Radiotherapy for oligometastatic tumor improved the prognosis of patients with non-small cell lung cancer (NSCLC). Thorac Cancer. 2019 May;10(5):1136-1140. doi: 10.1111/1759-7714.13054. Epub 2019 Apr 7. PMID 30957423
- [Background] Punnanitinont A, Kannisto ED, Matsuzaki J, Odunsi K, Yendamuri S, Singh AK, Patnaik SK. Sublethal Radiation Affects Antigen Processing and Presentation Genes to Enhance Immunogenicity of Cancer Cells. Int J Mol Sci. 2020 Apr 7;21(7):2573. doi: 10.3390/ijms21072573. PMID 32272797
- [Background] Shevtsov M, Sato H, Multhoff G, Shibata A. Novel Approaches to Improve the Efficacy of Immuno-Radiotherapy. Front Oncol. 2019 Mar 19;9:156. doi: 10.3389/fonc.2019.00156. eCollection 2019. PMID 30941308
- [Background] Bauml JM, Mick R, Ciunci C, Aggarwal C, Davis C, Evans T, Deshpande C, Miller L, Patel P, Alley E, Knepley C, Mutale F, Cohen RB, Langer CJ. Pembrolizumab After Completion of Locally Ablative Therapy for Oligometastatic Non-Small Cell Lung Cancer: A Phase 2 Trial. JAMA Oncol. 2019 Sep 1;5(9):1283-1290. doi: 10.1001/jamaoncol.2019.1449. PMID 31294762
- [Background] Theelen WSME, Peulen HMU, Lalezari F, van der Noort V, de Vries JF, Aerts JGJV, Dumoulin DW, Bahce I, Niemeijer AN, de Langen AJ, Monkhorst K, Baas P. Effect of Pembrolizumab After Stereotactic Body Radiotherapy vs Pembrolizumab Alone on Tumor Response in Patients With Advanced Non-Small Cell Lung Cancer: Results of the PEMBRO-RT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Sep 1;5(9):1276-1282. doi: 10.1001/jamaoncol.2019.1478. PMID 31294749
- [Background] Annede P, Cosset JM, Van Limbergen E, Deutsch E, Haie-Meder C, Chargari C. Radiobiology: Foundation and New Insights in Modeling Brachytherapy Effects. Semin Radiat Oncol. 2020 Jan;30(1):4-15. doi: 10.1016/j.semradonc.2019.08.009. PMID 31727299
- [Background] Gao S, Li N, Gao S, Xue Q, Ying J, Wang S, Tao X, Zhao J, Mao Y, Wang B, Shao K, Lei W, Wang D, Lv F, Zhao L, Zhang F, Zhao Z, Su K, Tan F, Gao Y, Sun N, Wu D, Yu Y, Ling Y, Wang Z, Duan C, Tang W, Zhang L, He S, Wu N, Wang J, He J. Neoadjuvant PD-1 inhibitor (Sintilimab) in NSCLC. J Thorac Oncol. 2020 May;15(5):816-826. doi: 10.1016/j.jtho.2020.01.017. Epub 2020 Feb 6. PMID 32036071